CLINICAL TRIAL: NCT02154555
Title: A Randomized Controlled Trial Evaluating Postoperative Debridement Following Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POD_001
Record Dates: First submitted 2014-04-25; First posted 2014-06-03 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Chronic Rhinosinusitis
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- no debridement (No Intervention): The postoperative clinical visits will occur at one week, one month, and three months following surgery. During all three postoperative visits, no debridement will be performed.
- debridement (Experimental): The postoperative clinical visits will occur at one week, one month, and three months following surgery. During the one week postoperative visit, the randomized unilateral debridement will be performed. Debridement includes removing any crust or mucous in the nose. During the one month and three month visit, the PI will only examine the nose.
  Interventions: Procedure: debridement

INTERVENTIONS:
Procedure: debridement — post-operative debridement at 1 week follow-up visit
  Arms: debridement

SUMMARY:
Chronic rhinosinusitis (CRS) is a common sinus and nasal condition affecting more than 33 million Americans. The treatment of CRS typically begins with maximal medical therapy however, when this fails to improve patient symptoms, surgical intervention is considered. Endoscopic sinus surgery (ESS) is a well-established treatment for refractory CRS with approximately 600,000 sinus surgeries performed annually in the United States alone. Despite the success of this intervention, up to 26% of patients experience complications following surgery, including middle meatal (MM) synechiae, edema, polyp recurrence, and middle turbinate lateralization. Currently, there is no consensus as to the postoperative care regime that is most effective at minimizing or preventing these potential complications. Therefore there is need for further study into the role of debridement, examining patients undergoing endoscopic sinus surgery while concurrently addressing the potential confounders of maximal medical therapies in the postoperative setting.

This prospective, randomized, single-blind, controlled study design will investigate the efficacy of postoperative debridement following ESS. Patients who have undergone ESS will have one nare randomized to debridement and the other to no debridement at the first week post-operative visit. In this way, the patients will act as their own controls in order to account for inter-patient variability in disease severity. The primary outcome will assess synechiae formation attributed to ESS. Secondary outcomes will include pain (side-specific) attributed to the debridement procedure as well as comparing pre and post endoscopy scores and SNOT-22 questionnaire responses.

DETAILED DESCRIPTION:
The significant heterogeneity present in the current literature regarding the use of postoperative debridement warrants additional studies that document postoperative protocols and use universally accepted endoscopy scores in order to consistently track patient outcomes. Further investigation into the efficacy of postoperative debridement is especially interesting with the potential benefits of further reduced synechiae formation and edema. Conversely, if objective evidence fails to demonstrate benefit of postoperative debridement, there could be significant cost and time saving for healthcare professionals in removing this therapy from the postoperative protocols.

We hypothesize that postoperative debridement will have a significant effect on reducing the rates of synechiae formation. In addition, we hypothesize that this improvement in synechiae development will also be matched by improvements in postoperative endoscopic sinus scoring, and patient's overall symptoms at 1 and 3 months postoperatively.

This study can clarify the efficacy of postoperative debridement and the potential benefits of further reduced synechiae formation and edema, and thus decrease the rates of complication and revision surgery. Conversely, if objective evidence fails to demonstrate benefit of postoperative debridement, there could be significant cost and time saving for healthcare professionals in removing this therapy from the postoperative protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Chronic Rhinosinusitis (as defined by the American Academy of Otolaryngology - Head & Neck Surgery)
* Consented to proceed with bilateral ESS
* Require bilateral middle meatus spacers postoperatively
* Adequate fluency in English to provide consent and complete surveys

Exclusion Criteria:

* History of immune deficiency
* Allergic fungal sinusitis
* Cystic Fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of synechiae - binary rating | 1 week, 1 month, and 3 months after surgery
  adhesions, scarring between middle turbinate and lateral nasal wall

SECONDARY OUTCOMES:
Change of Lund-Kennedy endoscopy score | before surgery at clinical visit when consent for surgery is obtained (within 9 month period before surgery)
Change of pain score - 10-point Likert scale | 1 week after surgery
  rated for each sinonasal cavity
Change of SNOT-22 score | before surgery at clinical visit when consent for surgery is obtained (within 9 month period before surgery)
  22-item sinonasal outcome test (SNOT-22) questionnaire score
10-point Likert scale | 1 month after surgery
  rated for each sinonasal cavity
pain score - 10-point Likert scale | 3 months after surgery
  rated for each sinonasal cavity
Lund-Kennedy endoscopy score | 1 week after surgery
Lund-Kennedy endoscopy score | 1 month after surgery
Lund-Kennedy endoscopy score | 3 months after surgery
SNOT-22 score | 1 week after surgery
  22-item sinonasal outcome test (SNOT-22) questionnaire score
SNOT-22 score | 1 month after surgery
  22-item sinonasal outcome test (SNOT-22) questionnaire score
SNOT-22 score | 3 months after surgery
  22-item sinonasal outcome test (SNOT-22) questionnaire score
pain score - 10-point Likert scale | before surgery at clinical visit when consent for surgery is obtained (within 9 month period before surgery)
  rated for each sinonasal cavity

CONTACTS AND LOCATIONS:
Overall Officials: John Lee, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No